CLINICAL TRIAL: NCT07058246
Title: Effectiveness of Mime Therapy and Conventional Therapy for the Patients of Bell's Palsy
Brief Title: Effectiveness of Mime Therapy vs Conventional Therapy for Bell's Palsy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Elite College of Management Sciences, Gujranwala, Pakistan (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2020-GCUF-079255
Record Dates: First submitted 2025-05-30; First posted 2025-07-10 (Actual); Last update posted 2025-07-10 (Actual); Status verified 2025-07

CONDITIONS: Bell Palsy
Keywords: Bell Palsy; Rehabilitation
MeSH Terms: conditions — Bell Palsy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental): Group A is the experimental group having 17 participants randomly chosen by using coin toss method according to inclusion and exclusion criteria.
  Baseline Treatment include DL2 electric stimulation at 20-50Hz for 90 repetitions and Infrared lamp placed 30-45cm away from the body for 10-15 minutes.
  Mime Therapy along with Conventional Therapy.
  Interventions: Other: Mime therapy with Conventional therapy
- Group B (Active Comparator): Group B is the active comparator group having 17 participants randomly chosen by using coin toss method according to inclusion and exclusion criteria.
  Baseline Treatment include DL2 electric stimulation at 20-50Hz for 90 repetitions and Infrared lamp placed 30-45cm away from the body for 10-15 minutes.
  Conventional Therapy.
  Interventions: Other: Conventional therapy

INTERVENTIONS:
Other: Mime therapy with Conventional therapy — Experimental group was given mime therapy along with conventional therapy. Mirror therapy, Raising eyebrows as if surprised, Widening eyes in shock, blinking rapidly, Extreme smiling, Eye closure with dramatic expressions, exaggeration nose wrinkling. pouting and mouth opening, expression transitions.
  Total sessions given are 4-5 per week in 3 weeks consist of 45 mins.
  Number of repetitions are 5-10 with the hold of 5 second x 2 sets.
  Arms: Group A
Other: Conventional therapy — Raising and lowering eyebrows, Wrinkling nose, smiling, frowning, massage.
  Total sessions given are 4-5 per week in 3 weeks consist of 45 mins.
  Number of repetitions are 5-10 with the hold of 5 second x 2 sets.
  Arms: Group B

SUMMARY:
The objective of this study is to evaluate the effectiveness of mime therapy and conventional therapy for improving facial functional mobility and coordination.

DETAILED DESCRIPTION:
This will be a Randomized Controlled Trial (RCT). Sample will be taken using Non-Probability Convenient Sampling. Sample size of 34 participants that will be randomly allocated into two groups using a coin toss method. Group A (intervention group) will receive mime therapy along with conventional therapy, while Group B (control group) will receive only conventional therapy were given 45 minutes per day for 3-4 sessions in a week for 3 weeks. Outcomes will be measured by using the Sunnybrook Facial Grading System for checking facial symmetry and the House-Brackmann Facial Grading System for measuring severity of paresis.

ELIGIBILITY:
Inclusion Criteria:

* Patient diagnosed with acute bell's palsy
* All genders and intact taste sensations
* No other neurological deficit involving face

Exclusion Criteria:

* Uncontrolled hypertension
* Stroke patients
* Patient with mental and dental implants
* Patient with recurrent facial palsy
* Patient with tumors, congenital defects, open wound

Ages: 25 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 34 (Actual)
Dates: Start 2025-04-01 (Actual); Primary Completion 2025-06-01 (Actual); Study Completion 2025-07-01 (Actual)

PRIMARY OUTCOMES:
Facial Disability Index | 4 months
  it includes physical well being scale which consist of 5 questions with a 0-5 scoring and social functional scale which consist of 5 questions with a 1-6 scoring.

SECONDARY OUTCOMES:
House Brackmann Facial Grading Scale | 4 months
  It classifies facial nerve function into six grades, ranging from Grade 1(normal function) to Grade 6 (complete paralysis). It is widely used for assessing facial nerve recovery.

CONTACTS AND LOCATIONS:
Overall Officials: Rimza Safdar, DPT, Principal Investigator — Elite College of Management sciences
Locations (1):
- Al Raee Hospital, Gujranwala, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Beurskens CH, Heymans PG. Mime therapy improves facial symmetry in people with long-term facial nerve paresis: a randomised controlled trial. Aust J Physiother. 2006;52(3):177-83. doi: 10.1016/s0004-9514(06)70026-5. PMID 16942452
- See also: In 2025, Islam Hussain and M Samir conducted a systemic review and meta analysis in which He concluded the effectiveness of mime therapy in improving clinical and functional outcomes. — https://ijtau.journals.ekb.eg/article_427692.html